CLINICAL TRIAL: NCT05555498
Title: Virtual Reality for Anxiety and Pain Management During Oocyte Retrieval in IVF/ICSI Treatment
Acronym: VitRo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof. Velja Mijatovic, Professor Doctor, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010170
Record Dates: First submitted 2022-03-04; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: IVF; Procedural Pain; Procedural Anxiety
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Masking Description: Patients are randomised between the intervention group where VR glasses are added to standard care with conscious sedation (intervention group), and the control group where only standard care consisting of conscious sedation (opioids with benzodiazepines) is applied. When assigned to the intervention group, the patient will wear VR-glasses during the entire procedure of oocyte retrieval in IVF/ICSI treatment. Due to the nature of the intervention, double blind randomisation is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: VR-glasses added to standard care of conscious sedation (Experimental): For the intervention group, Virtual Reality glasses will be administered on top of standard pain and anxiety management. Standard pain and management consists of conscious sedation, where benzodiazepines and opioids are administrered. In addition, participants are asked to complete 4 questionnaires on different times : immediately before, immediately after and three days after oocyte retrieval. In case of ongoing pregnancy, women are asked to complete a questionnaire approximately a month after their expected date of delivery.
  Interventions: Device: Virtual Reality glasses
- standard care consisting of conscious sedation (No Intervention): The control group will receive standard pain- and anxiety management during oocyte retrieval in IVF/ICSI treatment, consisting of opioids combined with benzodiazepines. This will result in a conscious sedated state. In addition, participants are asked to complete 4 questionnaires on different times : immediately before, immediately after and three days after oocyte retrieval. In case of ongoing pregnancy, women are asked to complete a questionnaire approximately a month after their expected date of delivery.

INTERVENTIONS:
Device: Virtual Reality glasses — The intervention used are Virtual Reality glasses. The VR-glasses used are designed by SyncVR medical (Utrecht, the Netherlands), and are applicable specifically for medical use. By distracting the patients' cognition from the procedure, using images and sounds, the patient hopefully experiences less pain and anxiety. Women can choose between relaxation excersises and nature films
  Arms: Intervention group: VR-glasses added to standard care of conscious sedation

SUMMARY:
Despite current anxiety and pain management during oocyte retrieval in IVF/ICSI treatment by conscious sedation, oocyte retrieval often remains painful and stressful for patients. An average pain score of 6.0 (expressed using VAS) and stress score of 41.63 (using STAI-S) were reported by previous researches. Previous research showed there might be a negative correlation between anxiety experienced in IVF/ICSI treatment, and ongoing pregnancy rate. Other researches nuance this. In addition, conscious sedation can give a variety of side effects such as apnea and respiratory depression.

The appliance of Virtual Reality is increasingly researched, in a variety of procedures. Previous researches showed that Virtual Reality was effective in the reduction of anxiety and pain experienced, also in the field of Gynaecology and Obstetrics. We hypothesized that Virtual Reality can aid in the reduction of anxiety and pain experienced during oocyte retrieval in IVF/ICSI treatment. We also aim to find a definitive answer on the question whether anxiety during IVF/ICSI treatment can negatively influence ongoing pregnancy rates.

DETAILED DESCRIPTION:
Patients undergoing oocyte retrieval as part of IVF/ICSI treatment are often still anxious and experience pain despite adequate management of both by applying conscious sedation, consisting of opioids combined with benzodiazepines. An average pain score of 6.0 during oocyte retrieval is reported by patients, expressed using the Visual Analogue Score (VAS). Very limited research has been done on anxiety experienced during oocyte retrieval by patients. However, in 2013 Turner et al. reported an average anxiety score of 41.63, objectified using the State-Trait Anxiety Inventory (STAI-S) of Spielberger et al. They also saw a higher pregnancy rate in women reporting a lower anxiety score (34.93 in pregnant women versus 44.35 in non-pregnant women, p=0.05). This finding was nuanced by other researches, they found no correlation between anxiety and IVF/ICSI outcomes.

There is an increased risk of side effects when benzodiazepines are added to opioids to induce conscious sedation. Due to the anxiolytic, sedative and amnesic effect of benzodiazepines, a reduction in anxiety experienced by patients is seen. Benzodiazepines combined with opioids additionally cause a depression of the central nervous system, resulting in a conscious sedative state. The patient is still fully conscious and able to communicate with the healthcare provider. However, the risk of respiratory side effects such as respiratory depression and apnea increases when conscious sedation is applied. No successful alternative to benzodiazepines has yet been found.

Virtual Reality is increasingly used successfully to reduce both anxiety and pain experienced by patients during a variety of procedures. Additionally, higher satisfaction scores by both the patient and care giver are reported when Virtual Reality was applied. By deriving the patient's cognition from the procedural pain using a Virtual Reality environment, subjective pain experienced by the patient is reduced. VR is increasingly used in the medical field, including in the field of Gynecology and Obstetrics. However, no studies have yet been conducted on the effectiveness of VR during oocyte retrieval.

Based on previous studies, where reduced pain and anxiety was seen when Virtual Reality was applied, we hypothesized that a VR intervention can aid in the reduction of pain and anxiety experienced by patients during oocyte retrieval. In addition, we hypothesize there is a higher ongoing pregnancy rate in women experiencing less anxiety during oocyte retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 43 years of age;
* Undergoing oocyte retrieval as part of IVF/ICSI treatment;
* Be able to understand and read the Dutch or English language.

Exclusion Criteria:

* Chronic use of pain medication;
* Chronic use of anti-depressants or sedatives;
* Women who previously underwent an oocyte retrieval with a VR intervention;
* Women undergoing oocyte retrieval because of fertility preservation;
* Women with visual or auditive impairment;
* Technology-related sensitivity such as motion-sickness, dizziness, epilepsy, seizures, active nausea and vomiting;
* Women who are not willing or able to give their informed consent.

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of anxiety during oocyte retrieval | 2 hours
  Assessed using the STAI-S. A score between 20 and 80 can be calculated. The higher the score, the more severe the anxiety experienced is.

SECONDARY OUTCOMES:
Reduction of pain scores during oocyte retrieval | 2 hours
  Measured using a VAS-score, scale 0-10. The higher the VAS-score, the more pain the participant exprienced.
Duration of the procedure | 2 hours
  When the patients' anxiety is reduced, it is expected that she is more relaxed and the procedure will run more smoothly resulting in a shorter duration of the procedure.
Satisfaction score of the patient | 2 hours
  Measured using the Numeric Rating Scale, with a scale from 0 to 10. The higher the NRS-score, the higher patient satisfaction.
satisfaction score of the care giver | 2 hours
  Measured using the Numeric Rating Scale, with a scale from 0 to 10. The higher the NRS-score, the higher care giver satisfaction.
Occurrence of side effects | 3 days
  Measured using a questionnaire, with a 5-point Likert Scale.
Ongoing pregnancy rate | 10 months
  Defined as the precence of a heart beat at 10 to 12 weeks gestation
Use of oral analgesics | 3 days
  Possible need for pain medication until 3 days after oocyte retrieval. Measured using a questionnaire that is send 3 days after oocyte retrieval.
Immersiveness in the VR program | 2 hours
  Measured using a questionnaire, with a 5-point Likert Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
No trial data will be shared with other researchers. Only the researchers involved in the trial will be able to see the data. All participants will be assigned an anonymous code. To this code, all study data will be collected. The key to the codes will be stored at the research center, in a sealed digital map.

REFERENCES:
- [Derived] van Haaps AP, Schreurs AMF, Rosielle K, Mijatovic V, Kallewaard JW, Dreyer K. No anxiety or pain reduction by Virtual Reality during oocyte retrieval in IVF/ICSI treatment: results of a randomized controlled trial. Hum Reprod. 2025 Oct 7:deaf193. doi: 10.1093/humrep/deaf193. Online ahead of print. PMID 41057042